CLINICAL TRIAL: NCT03986944
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Study to Assess the Efficacy and Safety of Linzagolix in Subjects With Moderate to Severe Endometriosis-associated Pain.
Brief Title: A Phase 3 Study to Confirm the Efficacy and Safety of Linzagolix to Treat Endometriosis-associated Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted due to the significant enrollment challenges encountered since its beginning. Screening and enrollment have been impacted by the COVID pandemic and more importantly by changes in the diagnosis and treatment of women with endometriosis.
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-OBE2109-002
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis
Keywords: Dysmenorrhea; Dyspareunia; Dyschezia; Non-menstrual pelvic pain
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Dyspareunia; Constipation | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Linzagolix 75 mg (Experimental)
  Interventions: Drug: 75 mg linzagolix tablet; Drug: Placebo tablet to match 200 mg linzagolix tablet; Drug: Placebo capsule to match Add-back capsule
- Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg) (Experimental)
  Interventions: Drug: 200 mg linzagolix tablet; Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg); Drug: Placebo tablet to match 75 mg linzagolix tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo tablet to match 75 mg linzagolix tablet; Drug: Placebo tablet to match 200 mg linzagolix tablet; Drug: Placebo capsule to match Add-back capsule

INTERVENTIONS:
Drug: 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg
Drug: 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg) — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo tablet to match 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg); Placebo
Drug: Placebo tablet to match 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg; Placebo
Drug: Placebo capsule to match Add-back capsule — For oral administration once daily
  Arms: Linzagolix 75 mg; Placebo

SUMMARY:
The primary objective of this study is to demonstrate the efficacy and safety of linzagolix administered orally once daily for 3 months at a dose of 75 mg alone or of 200 mg in combination with add-back hormone replacement therapy (ABT: estradiol (E2) 1 mg / norethisterone acetate (NETA) 0.5 mg) versus placebo, in the management of moderate to severe endometriosis-associated pain (EAP).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study to demonstrate the efficacy and safety of linzagolix administered orally once daily at doses of 75 mg alone and 200 mg in combination with low dose ABT (E2 1 mg/NETA 0.5 mg) versus placebo in the management of moderate to severe EAP in 450 women.

Eligible subjects who have completed the 6-month treatment period may enter a separate extension study for 6 additional months of active treatment (no placebo control). Subjects who do not continue in the extension study will enter a 6 month treatment-free follow-up phase.

ELIGIBILITY:
Key Inclusion Criteria:

The subject must have:

* Her most recent surgical and - if available - histological diagnosis of pelvic endometriosis up to 10 years before screening.
* Moderate to severe endometriosis-associated pain during the screening period.
* Regular menstrual cycles.
* BMI ≥ 18 kg/m2 at the screening visit.

Key Exclusion Criteria:

The subject will be excluded if she:

* Is pregnant or breast feeding or is planning a pregnancy within the duration of the treatment period of the study.
* Is less than 6 months postpartum or 3 months postabortion/ miscarriage at the time of entry into the screening period.
* Has had a surgical history of any major abdominal surgery within 6 months or any interventional surgery for endometriosis performed within a period of 2 months before screening.
* Did not respond to prior treatment with GnRH agonists or GnRH antagonists for endometriosis.
* Has a history of, or known, osteoporosis or other metabolic bone disease.
* Has chronic pelvic pain that is not caused by endometriosis and requires chronic analgesic or other chronic therapy which would interfere with the assessment of endometriosis-associated pain.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females Only
Enrollment: 85 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecomte, Study Director — ObsEva SA
Locations (112):
- United States (107):
  - Birmingham OBGYN / ID # 740, Birmingham, Alabama
  - Mesa Obstetricians and Gyneocologists / ID # 790, Mesa, Arizona
  - Precision Trials AZ, LLC / ID # 783, Phoenix, Arizona
  - Quality of LIfe Medical & Research Center, LLC / ID # 813, Tucson, Arizona
  - Visions Clinical Research-Tucson / ID # 754, Tucson, Arizona
  - Lynn Institute of the Ozarks / ID # 826, Little Rock, Arkansas
  - Applied Research Center of Arkansas / ID # 735, Little Rock, Arkansas
  - Join Clinical Trials / ID # 778, Huntington Park, California
  - Long Beach Clinical Trials, LLC / ID # 768, Long Beach, California
  - Matrix Clinical Research / ID # 751, Los Angeles, California
  - Futura Research, Org / ID # 781, Norwalk, California
  - National Research Institute / ID # 805, Panorama City, California
  - Precision Research Institute / ID # 792, San Diego, California
  - MD Strategies Research Centers / ID # 765, San Diego, California
  - Downtown Women's Health Care / ID # 718, Denver, Colorado
  - Center for Women's Health / ID # 761, Greenwood Village, Colorado
  - Physicians Research Options, LLC / Red Rocks Ob/Gyn / ID # 732, Lakewood, Colorado
  - Dr. David I. Lubetkin, LLC / ID # 703, Boca Raton, Florida
  - Helix Biomedics Clincial Research, LLC / ID # 750, Boynton Beach, Florida
  - Accel Research Sites, DeLand Clinical Research Unit / ID # 713, DeLand, Florida
  - Universal Axon Clinical Research / ID # 769, Doral, Florida
  - Clinical Neuroscience Solutions, Inc. / ID # 773, Jacksonville, Florida
  - South Florida Clinical Research Institute / ID # 747, Margate, Florida
  - Coral Way Research / ID # 799, Miami, Florida
  - Suncoast Research Group, LLC / ID # 756, Miami, Florida
  - Biotech Pharmaceutical Group LLC / ID # 786, Miami, Florida
  - La Salud Research Clinic, Inc. / ID # 824, Miami, Florida
  - Suncoast Research Associates, LLC / ID # 760, Miami, Florida
  - LCC Medical Research Institute / ID # 814, Miami, Florida
  - Global Health Research Center, Inc. / ID # 787, Miami Lakes, Florida
  - Sensible Healthcare / ID # 749, Ocoee, Florida
  - A Premier Medical Research of Florida, LLC / ID # 752, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc. / ID # 731, Orlando, Florida
  - Omega Research Orlando, LLC / ID # 785, Orlando, Florida
  - Clinical Associates of Orlando, LLC / ID # 779, Orlando, Florida
  - Synexus Clinical Research US, Inc. / ID # 725, Orlando, Florida
  - Physician Care Clinical Research LLC / ID # 810, Sarasota, Florida
  - University of South Florida / ID # 738, Tampa, Florida
  - GCP Clinical Research, LLC / ID # 825, Tampa, Florida
  - Atlanta Women's Research Institute, Inc. / ID # 727, Atlanta, Georgia
  - Sonara Clinical Research, LLC / ID # 720, Meridian, Idaho
  - Moore Health Wellness Research Institute, LLC / ID # 795, Chicago, Illinois
  - Providea Health Partners LLC / ID # 734, Evergreen Park, Illinois
  - Cypress Medical Research Center, LLC / ID # 755, Wichita, Kansas
  - Horizon Research Group of Opelousas, LLC / ID # 757, Eunice, Louisiana
  - Praetorian Pharmaceutical Research / ID # 739, Marrero, Louisiana
  - Women Under Study, LLC / ID # 820, New Orleans, Louisiana
  - Johns Hopkins University, School Of Medicine / ID # 816, Baltimore, Maryland
  - Pharmasite Research Inc / ID # 838, Baltimore, Maryland
  - Continental Clinical Solutions, LLC / ID # 777, Towson, Maryland
  - NECCR Fall River, LLC / Id # 712, Fall River, Massachusetts
  - Onyx Clinical Research / ID # 793, Flint, Michigan
  - CMEP/CMU health / ID # 812, Saginaw, Michigan
  - Valley OBGYN / ID # 704, Saginaw, Michigan
  - Saginaw Valley Medical Research Group, LLC / ID # 743, Saginaw, Michigan
  - Office of Edmond Pack, MD / Id # 818, Las Vegas, Nevada
  - Lawrence OB/GYN clinical Research, LLC / ID # 742, Lawrenceville, New Jersey
  - Albuquerque Clinical Trials, Inc. / ID # 707, Albuquerque, New Mexico
  - Carolina Institute for Clinical Research / ID # 728, Fayetteville, North Carolina
  - Unified Women's Clinical Research - Green Valley OBGYN / ID # 719, Greensboro, North Carolina
  - Eastern Carolina Women's Center / Id # 794, New Bern, North Carolina
  - Unified Women's Clinical Research - Raleigh / Id # 714, Raleigh, North Carolina
  - Carolina Medical Trials, LLC / ID # 788, Winston-Salem, North Carolina
  - ClinOhio Research Services, LLC / ID # 722, Columbus, Ohio
  - Complete Healthcare for Women / ID # 801, Columbus, Ohio
  - Wright State Physicians / ID # 733, Dayton, Ohio
  - Hilltop OBGYN / ID # 711, Franklin, Ohio
  - Oregon Health & Science University / ID # 791, Portland, Oregon
  - OB/GYN Associates of Erie / ID # 706, Erie, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center / ID # 804, Hershey, Pennsylvania
  - The Clinical Trial Center / ID # 744, Jenkintown, Pennsylvania
  - VitaLink Research - Upstate / ID # 789, Greenville, South Carolina
  - Clinical Trials of South Carolina / ID # 741, North Charleston, South Carolina
  - VitaLink Research Spartanburg / ID # 753, Spartanburg, South Carolina
  - Seasons at Bristol / ID # 705, Bristol, Tennessee
  - WR-ClinSearch, LLC / ID # 821, Chattanooga, Tennessee
  - University of Tennessee Medical Center / ID # 780, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc / ID # 772, Memphis, Tennessee
  - Clinical Research Associates Inc / ID # 802, Nashville, Tennessee
  - Women Partners in Health / ID # 836, Austin, Texas
  - Austin Area ObGyn PLLC / ID # 701, Austin, Texas
  - Christina Sebestyen MD, P.A. dba OBGYN North / ID # 764, Austin, Texas
  - Christus St. Elizabeth Gadolin Research, LLC / ID # 774, Beaumont, Texas
  - HCWC dba DiscoveryClinical Trials / ID # 771, Dallas, Texas
  - UT Southwestern Medical Center / ID # 823, Dallas, Texas
  - Signature Gyn Services / ID # 726, Fort Worth, Texas
  - Georgetown OB/GYN / ID # 770, Georgetown, Texas
  - Ventavia Research Group, LLC / ID # 729, Houston, Texas
  - Vilo Research Group / ID # 709, Houston, Texas
  - UT Health Clinical Res Ctr / ID # 828, Houston, Texas
  - TMC Life Research, Inc. / ID # 809, Houston, Texas
  - MacArthur OB-Gyn Research / ID # 840, Irving, Texas
  - Medical Colleagues of Texas / ID # 819, Katy, Texas
  - FMC Science / ID # 730, Lampasas, Texas
  - Maximos OB/GYN / ID # 737, League City, Texas
  - DCT-McAllen Primary Care Research, LLC dba Discovery Clinical Trials / ID # 803, McAllen, Texas
  - DCT-AACT, LLC dba Discovery Clinical Trials / ID # 815, Pflugerville, Texas
  - Northeast Clinical Research of San Antonio, LLC / ID # 710, Schertz, Texas
  - Physicians Research Options PRO / ID # 766, Draper, Utah
  - Physicians' Res Options - PG / ID # 833, Pleasant Grove, Utah
  - Wasatch Clinical Research / ID # 746, Salt Lake City, Utah
  - Highland Clinical Research / ID # 708, Salt Lake City, Utah
  - Clinical Research Partners, LLC / ID # 715, Richmond, Virginia
  - Clinical Research Partners, LLC / ID # 775, Richmond, Virginia
  - Tidewater Clinical Research The Group for Women / ID # 716, Virginia Beach, Virginia
  - Seattle Women's: Health, Research, Gynecology / ID # 702, Seattle, Washington
  - Seattle Reproductive Medicine / ID # 811, Seattle, Washington
- Canada (3):
  - CARe Clinic / ID # 872, Red Deer, Alberta
  - McMaster University Medical Centre / ID # 870, Hamilton, Ontario
  - Victory Reproductive Care / ID # 873, Windsor, Ontario
- Puerto Rico (2):
  - Ponce Medical SChool Foundation Inc./ CAIMED Center / ID # 891, Ponce
  - Puerto Rico Medical Research Inc. / ID # 890, Ponce

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 492 subjects screened, 85 were randomized. Between randomization and Day 1 (i.e., first day of dosing), 1 subject in the placebo group discontinued due to protocol deviation. Thus, 84 randomized subjects were treated and comprised the Safety Analysis Set.
Pre-assignment Details: Participants with a diagnosis of pelvic endometriosis were enrolled in a 1:1:1 ratio in one of three treatment groups: LGX 75 mg, LGX 200 mg+ABT or Placebo.
Groups:
- LGX 75 mg: One Linzagolix 75 mg tablet, one Linzagolix 200 mg matching placebo tablet and one ABT matching placebo capsule were administered once daily orally for 6 months.
- LGX 200 mg+ABT: One Linzagolix 200 mg tablet and one Linzagolix 75 mg matching placebo tablet and ABT capsules (E2 1 mg / NETA 0.5 mg) were administered once daily orally for 6 months.
- Placebo: One Linzagolix 75 mg matching placebo tablet one Linzagolix 200 mg matching placebo tablet and ABT matching placebo capsule were administered once daily orally for 6 months.
Period: Overall Study
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
Started | 28 | 29 | 27
Completed | 13 | 10 | 8
Not Completed | 15 | 19 | 19
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 5
Not completed — Study termination | 10 | 10 | 10
Not completed — Discontinuation after moving to Follow-up Period [Study termination per Sponsor] | 1 | 0 | 0
Not completed — Discontinuation after moving to Follow-up Period [Subject's Request (Family Issue)] | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Amongst the 85 randomized subjects, 84 subjects were included in the safety analysis set (1 subject in the placebo group discontinued due to protocol deviation).
Groups:
- Total: Total of all reporting groups
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 27 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 27 | 84
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (7.2) | 33.4 (6.4) | 32.1 (6.9) | 32.7 (6.8)
Age, Customized [Median (Inter-Quartile Range); unit: years] | 32.5 [28.0 to 36.0] | 34.0 [29.0 to 37.0] | 31.0 [26.0 to 37.0] | 33.0 [28.0 to 37.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 27 | 84
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 12 | 9 | 28
  Not Hispanic or Latino | 20 | 17 | 18 | 55
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 5 | 10
  White | 22 | 27 | 20 | 69
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 0 | 3
  Puerto Rico | 4 | 2 | 0 | 6
  United States | 23 | 25 | 28 | 76
Weight [Mean (Standard Deviation); unit: kg] | 78.130 (16.904) | 76.540 (20.207) | 71.280 (16.050) | 75.379 (17.885)
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.08 (5.57) | 28.54 (8.48) | 26.61 (5.84) | 28.10 (6.79)

OUTCOME MEASURES:

1. Primary Outcome: Dysmenorrhea
Description: Change at Month 3 from baseline in the mean daily assessment of dysmenorrhea (DYS) measured on a 4-point Verbal Rating Scale (VRS) using an electronicdiary
  * The 4-point VRS scale for DYS ranges from 0 to 3 (0: No pain; 1: Mild pain; 2: Moderate pain; 3: Severe pain).
  * A negative change in scores would be indicative of an improvement in the pain of DYS.
Time Frame: Baseline to Month 3
Population: Due to the COVID-19 pandemic, the study was terminated early and only 85 out of the planned 450 subjects were randomized. As there were insufficient number of treated subjects at study termination, no analyses of efficacy were conducted. This time, we calculated mean±SD from only 6 subjects with DYS & NMPP data on both D1 & M3 and entered them as efficacy results in this table. There were no other subjects besides these 6 who had both data at baseline and another time point (M3, M6, M9 or M12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
Number analyzed (Participants) | 2 | 2 | 2
score on a scale | -0.5 (0.5) | 0.0 (0.0) | 0.5 (0.5)

2. Primary Outcome: Non-menstrual Pelvic Pain
Description: Change at Month 3 from baseline in the mean daily assessment of non-menstrual pelvic pain (NMPP) measured on a 4-point Verbal Rating Scale (VRS) using anelectronic diary
  * The 4-point VRS scale for NMPP ranges from 0 to 3 (0: No pain; 1: Mild pain; 2: Moderate pain; 3: Severe pain).
  * A negative change in scores would be indicative of an improvement in the NMPP.
Time Frame: Baseline to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
Number analyzed (Participants) | 2 | 2 | 2
score on a scale | -1.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: - Treatment Period: 6 months (Day 1 to Month 6) - Follow-up Period: 6 months (Month 6 to Month 6 FU)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial subject administered an investigational medicinal product (IMP) and which did not necessarily have a causal relationship with this treatment. Therefore, AE was any unfavourable sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP.
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 10/28 | 16/29 | 12/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=28) | LGX 200 mg+ABT (N=29) | Placebo (N=27)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
In this study, two co-primary endpoints, 1) clinically meaningful reduction up to Month 3 and 2) a stable/decreased use of analgesics for EAP of DYS & NMPP, were planned. Although the Responder Threshold Analysis was needed to evaluate the effectiveness of reducing pain, the clinical-meaningful response threshold couldn't be calculated due to the early study termination and the low number of subjects randomized. So, we showed the limited data of the changes up to Month 3 in DYS & NMPP instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT03986944/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03986944/SAP_003.pdf